CLINICAL TRIAL: NCT06855173
Title: Active External Rewarming from Accidental Hypothermia - a Dose-response Pilot Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/855256
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Accidental Hypothermia
Keywords: hypothermia; active external rewarming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- One active external rewarming device (Experimental): Participants in this group will recieve one active external rewarming device
  Interventions: Device: Active external rewarming device
- Two active external rewarming devices (Experimental): Participants in this group will recieve two active external rewarming devices
  Interventions: Device: Active external rewarming device; Device: Active external rewarming device 2
- Four active external rewarming devices (Experimental): Participants in this group will recieve four active external rewarming devices
  Interventions: Device: Active external rewarming device; Device: Active external rewarming device 2; Device: Active external rewarming device 3; Device: Active external rewarming device 4

INTERVENTIONS:
Device: Active external rewarming device — Electrical heating blanket
Device: Active external rewarming device 2 — Electrical heating blanket
  Arms: Four active external rewarming devices; Two active external rewarming devices
Device: Active external rewarming device 3 — Electric heating blanket
  Arms: Four active external rewarming devices
Device: Active external rewarming device 4 — Electric heating blanket
  Arms: Four active external rewarming devices

SUMMARY:
The aim of this pilot study is to evaluate if there is a dose-response relationship between the use of active external rewarming devices and core temperature rewarming rate from simulated accidental hypothermia. Volunteer research participants will be cooled in a field laboratory, and they will recieve medications to inhibit shivering, enabeling a drop in core temperature. Subsequently, they will be treated with either one, two or four heating blankets, and analyses will be performed to investigate whether we are able to find a difference between the three groups.

DETAILED DESCRIPTION:
The aim of this pilot study is to evaluate if there is a dose-response relationship between the use of active external rewarming devices and core temperature rewarming rate from simulated accidental hypothermia. Volunteer research participants will be cooled in a field laboratory, and they will recieve medications to inhibit shivering, enabeling a drop in core temperature. All participants will be monitored extensively using a trans-nasal esophageal temperature probe, ECG, SpO2, Blood pressure, skin temperature and with subjective scores. After the cooling phase, the participants will be treated with either one, two or four heating blankets assigned in a randomized order, and analyses will be performed to investigate whether we are able to find a difference between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Normal BMI
* Smoking

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-11 (Estimated); Primary Completion 2025-03-12 (Estimated); Study Completion 2025-03-12 (Estimated)

PRIMARY OUTCOMES:
Esophageal temperature rewarming rate | 1 hour
  Developement of esophageal temperature during the rewarming phase after cooling. Participants will be shiver-inhibited in this phase of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Thomassen, MD, PhD, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Risk of identifiable data due to a low number of participants